CLINICAL TRIAL: NCT00580047
Title: Effects of Zoledronic Acid Versus Alendronate on Bone Loss After Kidney and Kidney/Pancreas Transplant
Brief Title: Effects of Zoledronic Acid Versus Alendronate on Bone Loss After Kidney and Kidney/Pancreas Transplants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0437-02-FB
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Renal Insufficiency
Keywords: bone density; osteopenia; transplant; zoledronic acid; alendronate
MeSH Terms: conditions — Renal Insufficiency; Bone Diseases, Metabolic | interventions — Zoledronic Acid; Calcium; Vitamin D; Calcium Citrate; Calcium Carbonate; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 Zoledronic Acid (Active Comparator): Zoledronic Acid 4mg intravenously once a year for 2 years
  Interventions: Drug: Zoledronic Acid
- 2 Alendronate (Active Comparator): Alendronate 70mg orally once a week for 2 years
  Interventions: Drug: Alendronate
- 3 Placebo (Placebo Comparator): Combination drug entity: calcium 1200 mg with vitamin D 800 International Units daily
  Interventions: Combination Product: Calcium with vitamin D

INTERVENTIONS:
Drug: Zoledronic Acid — 4mg IV Annually
  Other Names: Zometa
  Arms: 1 Zoledronic Acid
Combination Product: Calcium with vitamin D — 1200 mg Calcium with 800 International Units of vitamin D
  Other Names: calcium citrate; calcium carbonate
  Arms: 3 Placebo
Drug: Alendronate — 70mg weekly
  Other Names: Fosamax
  Arms: 2 Alendronate

SUMMARY:
The study is designed to look at the effect of different bone treatment plans on bone loss after kidney or kidney/pancreas transplant.

DETAILED DESCRIPTION:
The aims are to determine baseline bone mineral density (BMD) in kidney and kidney/pancreas transplant patients who will be randomized to weekly alendronate, annual zoledronic acid infusions or placebo (calcium with Vitamin D). These patients will be followed for two years with annual bone density testing as well as biochemical markers. A secondary aim is to evaluate the compliance.

ELIGIBILITY:
Inclusion Criteria:

* Transplant patients who have had a kidney or kidney/pancreas transplant in the last 150 days with adequate kidney function as defined by a calculated creatine clearance of 35ml/min or more and serum creatinine less than 3.0

Exclusion Criteria:

* Dual X-ray Absorptiometry (DXA) T-score at the spine or hip of -3 or lower
* History of more than one vertebral or non-vertebral fracture in the past two years
* Abnormalities of the esophagus which delay esophageal emptying
* Inability to stay upright for 30 minutes
* Pregnant, nursing women or women not using an effective form of birth control
* Hypocalcemia
* Hypercalcemia
* Calculated creatinine clearance of <35 ml/min or serum creatinine > 3.0
* Patients already treated with bisphosphonates within the past one year
* Patients unable to undergo DXA
* Patients with cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-12-01 (Actual); Primary Completion 2014-07-29 (Actual); Study Completion 2014-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Mack, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Yao M, Xu JH, Shu B, Wang YJ, Cui XJ. Bisphosphonates for prevention of osteopenia in kidney-transplant recipients: a systematic review of randomized controlled trials. Osteoporos Int. 2016 May;27(5):1683-90. doi: 10.1007/s00198-015-3465-7. Epub 2016 Jan 5. PMID 26733377
- [Background] Shane E, Cohen A, Stein EM, McMahon DJ, Zhang C, Young P, Pandit K, Staron RB, Verna EC, Brown R, Restaino S, Mancini D. Zoledronic acid versus alendronate for the prevention of bone loss after heart or liver transplantation. J Clin Endocrinol Metab. 2012 Dec;97(12):4481-90. doi: 10.1210/jc.2012-2804. Epub 2012 Sep 28. PMID 23024190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients from the Kidney Pancreas Transplant clinic at the University of Nebraska Medical Center who underwent a kidney, pancreas, or kidney-pancreas transplant from 2003 to 2009 were invited to participate.
Pre-assignment Details: Participants were recruited during the transplant hospitalization or within 30 days of transplantation. They were excluded if they had an esophageal abnormality, bone density T-score of -3 or lower, fracture in the last 2 years, Cr Cl of 35 or less, inability to sit upright for 30 minutes after swallowing a medication.
Groups:
- Intravenous Bisphosphonate Post Transplantation: Zoledronic Acid 4mg
  Zoledronic Acid: 4mg IV Annually
- Oral Bisphosphonate Post Transplantation: Alendronate 70mg
  Alendronate: 70mg weekly
- Placebo Group Post Transplantation: Calcium 1200mg Vitamin D 800IU
  calcium and Vitamin D: 1200 mg Calcium 800 International Units Vitamin D
Period: Overall Study
Arm/Group | Intravenous Bisphosphonate Post Transplantation | Oral Bisphosphonate Post Transplantation | Placebo Group Post Transplantation
Started | 24 | 23 | 12
Completed | 21 | 21 | 10
Not Completed | 3 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Men and women post kidney or kidney pancreas transplantation
Groups:
- Oral Bisphosphonate Post Tranpslantation: Alendronate 70mg
  Alendronate: 70mg weekly
- Placebo Post Transplantation: Calcium 1200mg Vitamin D 800IU
  calcium and Vitamin D: 1200 mg Calcium 800 International Units Vitamin D
- Total: Total of all reporting groups
Arm/Group | Intravenous Bisphosphonate Post Transplantation | Oral Bisphosphonate Post Tranpslantation | Placebo Post Transplantation | Total
Number analyzed (Participants) | 24 | 23 | 12 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11) | 50 (15) | 46 (12) | 47 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 2 | 20
  Male | 13 | 16 | 10 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 12 | 59
Spine bone density [Mean (Standard Deviation); unit: grams/cm2] — mean spine bone density in g/cm2
  grams/cm2 | 1.5 (0.03) | 1.28 (0.046) | 1.12 (0.05) | 1.3 (.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Posterior Anterior (PA) Spine Bone Density From Baseline to 24 Months Post Transplant
Description: Posterior Anterior (PA) spine bone density was measured by dual energy x-ray absorptiometry (DXA) at baseline and 24 months post transplant. The percentage change in the PA spine bone density was then compared from baseline to 24 months post transplant.
Time Frame: 24 months
Population: Percentage change in spine bone density from baseline to 24 months
Measure: Number; unit: percentage of change of bone density
Groups:
- Intravenous Bisphosphonate Post Transplantation: Zoledronic Acid 4mg
  Zoledronic Acid: 4mg IV Annually
  8% increase
- Oral Bisphosphonate Post Transplantation: Alendronate 70mg
  Alendronate: 70mg weekly
  8% increase
- Placebo Group Post Transplantation: Calcium 1200mg Vitamin D 800IU
  calcium and Vitamin D: 1200 mg Calcium 800 International Units Vitamin D
  8% increase
Arm/Group | Intravenous Bisphosphonate Post Transplantation | Oral Bisphosphonate Post Transplantation | Placebo Group Post Transplantation
Number analyzed (Participants) | 24 | 23 | 12
percentage of change of bone density | 8.1 | 6.6 | 6.5

2. Secondary Outcome: Compliance With Zoledronic Acid, Alendronate and/or Calcium/Vitamin D Supplementation
Description: Compare compliance where a study coordinator interviewed patients as to how often they missed the once a week oral alendronate, missed taking calcium and vitamin D supplementation, or missed the once a year IV Reclast.
Time Frame: 24 months
Population: Compliance in study arm
Measure: Number; unit: percentage of compliance
Groups:
- Intravenous Bisphosphonate Post Transplantation: Zoledronic Acid 4mg
  Zoledronic Acid: 4mg IV Annually
  7.9% increase in spine bone density
- Oral Bisphosphonate Post Transplantation: Alendronate 70mg
  Alendronate: 70mg weekly
  5.8% increase in spine bone density
- Placebo Group Post Transplantation: Calcium 1200mg Vitamin D 800IU
  calcium and Vitamin D: 1200 mg Calcium 800 International Units Vitamin D
  6.2% increase in spine bone density
Arm/Group | Intravenous Bisphosphonate Post Transplantation | Oral Bisphosphonate Post Transplantation | Placebo Group Post Transplantation
Number analyzed (Participants) | 24 | 23 | 12
percentage of compliance | 100 | 80 | 80
Statistical Analysis 1: Comparison: Intravenous Bisphosphonate Post Transplantation vs Oral Bisphosphonate Post Transplantation; Test type: Other; The intervention groups were compared for compliance to either having annual IV zoledronic acid, taking weekly oral alendronate, and taking calcium/vitamin D supplementation

ADVERSE EVENTS:
Time Frame: 2 years
Description: A study coordinator helped the patient complete a questionnaire of potential side effects/adverse events
Groups:
- Intravenous Bisphosphonate After Tranpslant: Zoledronic Acid 4mg
  Zoledronic Acid: 4mg IV Annually
- Oral Bisphosphonate After Transplant: Alendronate 70mg
  Alendronate: 70mg weekly
- Placebo After Transplant: Calcium 1200mg Vitamin D 800IU
  calcium and Vitamin D: 1200 mg Calcium 800 International Units Vitamin D
Arm/Group | Intravenous Bisphosphonate After Tranpslant | Oral Bisphosphonate After Transplant | Placebo After Transplant
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/12
Other Adverse Events (participants affected / at risk) | 2/24 | 4/23 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Bisphosphonate After Tranpslant (N=24) | Oral Bisphosphonate After Transplant (N=23) | Placebo After Transplant (N=12)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample sizes and missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No